CLINICAL TRIAL: NCT01808885
Title: A 24-Week, Ph1b, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study, to Assess the Safety Profile of Olesoxime in Patients With Stable Relapsing Remitting Multiple Sclerosis Treated With Interferon Beta.
Brief Title: Safety Study of Olesoxime in Patients With Stable Relapsing Remitting Multiple Sclerosis Treated With Interferon Beta.
Acronym: MSREPAIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Hôpital de la Timone (Other); SGS S.A. (Industry); STRAGEN Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WP29866; 2012-005186-12 (EudraCT Number); TRO19622CLEQ1585-1 (Other: trophos id)
Record Dates: First submitted 2013-02-12; First posted 2013-03-11 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: safety; multiple sclerosis; olesoxime; double-blind; randomized
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — olesoxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- olesoxime (TRO19622) (Experimental): olesoxime (3 caps: 495 mg, od) will be administered orally as 165 mg soft capsules for 6 months.
  Investigational products will be allocated in a 1:1 ratio from Baseline/Visit 0 to Week 24 (Visit 3/Final Visit).
  Interventions: Drug: olesoxime (TRO19622)
- placebo (Placebo Comparator): placebo (3 soft capsules, od) will be administered orally for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olesoxime (TRO19622) — olesoxime (3 caps: 495 mg, od) will be administered orally as 165 mg soft capsules for 6 months.
  Investigational products will be allocated in a 1:1 ratio from Baseline/Visit 0 to Week 24 (Visit 3/Final Visit).
  Other Names: TRO19622 (olesoxime)
  Arms: olesoxime (TRO19622)
Drug: placebo — placebo capsule shells with identical appearance as the active compound TRO19622
  Arms: placebo

SUMMARY:
This is a 24-week phase 1b, randomized, double-blind, placebo-controlled, parallel-group, multicenter safety study comparing the tolerance profile of olesoxime (495 mg, od) when administered on top of Interferon beta in patients with stable Relapsing Remitting Multiple Sclerosis. Patients will be randomly allocated to olesoxime (495 mg, od) or placebo in a 1:1 ratio.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the general safety and tolerability of olesoxime (495 mg, od), compared to placebo when administered in combination with Interferon beta over a 24-week treatment period in patients with stable Relapsing Remitting Multiple Sclerosis.

The secondary objective of this study is to evaluate the feasibility of multicenter protocols for measurement of neurodegeneration and remyelination by MRI as well as the plasma exposure to olesoxime (495 mg, od).

MRI will be performed to all patients to assess effects of olesoxime on brain inflammation as well as to assess measures of brain atrophy, neuronal damage and myelination status at Baseline, 12 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* Diagnosed with Relapsing Remitting Multiple Sclerosis. Patients must be stable defined as free from relapsing episode for at least 6 months prior to Baseline
* Patients must be treated with Interferon beta for at least one year
* Patients must have an Expanded Disability Status Scale (EDSS) score ≤ 5
* Female patients must be post-menopausal (defined as at least 12 months post cessation of menses), surgically sterile or, if of childbearing potential, using a reliable method of contraception for at least 3 months prior to Baseline and during the study. In addition, female patients must not be lactating
* Patients must be able to understand and comply with study requirements
* Patients must provide a written, dated and signed informed consent prior to any study procedure

Exclusion Criteria:

* Any relapse of multiple sclerosis within the past 6 months prior to Screening Visit/Visit -1
* Any change in Interferon treatment within the past year prior to Screening Visit (Visit -1)
* Expected use of another disease modifying therapy from Screening Visit/Visit -1 to Visit 3/Final Visit
* Patients unable to undergo MRI scan
* Current or expected use of a medication that could interfere with olesoxime pharmacology (e.g. tamoxifen)
* Current or expected use of lipid lowering agents (ezetimibe, bile salt chelators, fibrates, phytosterols) other than statins
* Known hypersensitivity to olesoxime or any of its components
* History of alcohol or drug abuse within the last 6 months, or addiction within the last 2 years prior to Baseline Visit
* Positive urinary pregnancy test at Baseline Visit
* History of hepatitis B/C or HIV positive serology
* Hepatic impairment (aspartate aminotransferase (AST) and alanine aminotransferase (ALT)> 3 × ULN) at Baseline Visit
* History of renal impairment defined by a serum creatinine value > 176 μmol/L (2.0 mg/dL) at Baseline Visit
* Abnormal and clinically significant ECG at Screening Visit/Visit -1 as assessed by a cardiologist
* Current or expected use of oral or intramuscular corticosteroids within 3 months prior to the Screening Visit. Only stable dose regimens of inhaled and topical corticosteroids are allowed during the study
* History of any clinically relevant gastrointestinal (GI), respiratory, psychiatric, neurological, kidney, liver, cardiac diseases, bleeding disorder, other disease/condition or abnormal physical finding which may interfere with the study objectives or put the patient's safety at risk, as judged by the Investigator
* Patients with an active chronic disease (or stable but treated with immune therapy) of the immune system other than Multiple Sclerosis (MS)
* History of malignancy of any organ, treated or non-treated within the past 5 years
* Current participation or participation within 30 days prior to study entry, in another investigational drug or device study, or previous enrolment in the present study
* Any direct involvement with the study conduct at site or any family link with study site staff
* Pregnant, parturient or lactating women, as per Public Health Code (CSP)(Article L-1121-5)
* Persons deprived of their liberty by a judicial or administrative decision, and those admitted to a health or social facility, as per CSP (Article L-1121-6)
* Persons covered by a measure of legal protection or unable to provide a written, dated and signed informed consent, as per CSP(Article L-1121-8)
* Patient without Social Security Insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Safety criteria | The primary endpoint of this study will be the cumulative incidence of AE/SAE assessed by ongoing monitoring at week 24 (day 168)
  Cumulative incidence of adverse events/serious adverse events (i.e. total number per patient) as assessed by ongoing monitoring.

SECONDARY OUTCOMES:
MRI Parameters | Baseline (Visit 0), Week 12 (Visit 2) and Week 24 (Visit 3/Final Visit)
  1. Number of Gadolinium-enhancing lesions on T1-weighted images
  2. Number of new or enlarged lesions on T2-weighted images

OTHER OUTCOMES:
Exploratory MRI Parameters | Baseline (Visit 0), Week 12 (Visit 2) and Week 24 (Visit 3/Final Visit)
  Exploratory Endpoints:
  The following parameters will be assessed in terms of feasibility and reproducibility in a multicenter setting:
  3. Whole brain atrophy volume assessed by 3D-T1-weighted images. 4. Demyelination and remyelination processes assessed by Diffusion Tensor Imaging.
  5. Remyelination processes assessed by Magnetization Transfer Ratio. 6. Neuroaxonal damage assessed by sodium 23 imaging in one center.

CONTACTS AND LOCATIONS:
Overall Officials: Jean PELLETIER, MD, Principal Investigator — Head of Neurology Department, UMR CRMBM CNRS 6612, Timone University Hospital, Marseille, France; Ayman TOURBAH, MD, Principal Investigator — Professor of Neurology, Neurology Department & University of Reims; Gilles EDAN, MD, Principal Investigator — Professor of Clinical Neurology, Head of Neurology Department, Pontchaillou Hospital, Rennes, France
Locations (3):
- France (3):
  - Timone University Hospital, Neurology Department, UMR CRMBM CNRS 6612, Marseille
  - CHU Reims, Maison Blanche Hospital, Neurology Department & University of Reims, Reims
  - CHU Pontchaillou, Neurology Department, Rennes